CLINICAL TRIAL: NCT06056349
Title: An Open Label Benzodiazepine Study for the Treatment of Seizure Clusters in a Third Level Mexican Neurological Center
Brief Title: Benzodiazepine Study for the Treatment of Seizure Clusters in a Third Level Mexican Neurological Center
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: El Instituto Nacional de Neurologia y Neurocirugia Manuel Velasco Suarez (Other)
Responsible Party: Principal Investigator, Elma Paredes-Aragón, Staff Neurologist, Epileptologist, El Instituto Nacional de Neurologia y Neurocirugia Manuel Velasco Suarez
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05/23
Record Dates: First submitted 2023-04-25; First posted 2023-09-28 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Cluster Seizure
Keywords: seizure cluster; epilepsy; rescue medication; benzodiazepines
MeSH Terms: conditions — Epilepsy | interventions — Midazolam; Clonazepam

STUDY DESIGN:
Intervention Model Description: This is an open label, randomnized, prospective clinical trial, with a 1:1:1 aleatorization of a single third level specialized neurological center.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Orodispersable clonazepam (Experimental): 50 patients will receive oral orodispersable clonazepam.
  Interventions: Drug: ClonazePAM Oral Product
- Buccal midazolam (Experimental): 50 patients will receive buccal midazolam.
  Interventions: Drug: Midazolam oral solution
- Conventional treatment (Active Comparator): 50 patients will receive "usual/ conventional treatment of seizure clusters"
  Interventions: Other: Usual medication/ traditional

INTERVENTIONS:
Drug: Midazolam oral solution — Buccal administration
  Other Names: midazolam
  Arms: Buccal midazolam
Drug: ClonazePAM Oral Product — Orodispersable
  Other Names: clonazepam
  Arms: Orodispersable clonazepam
Other: Usual medication/ traditional — Medication that is usually used in the emergency department
  Arms: Conventional treatment

SUMMARY:
The aim of this study is to determine the efficacy in seizure reduction when comparing orodispersable clonazepam versus usual treatment (i.e. medication load, intravenous high- dose benzodiazepines) of seizure clusters in a third level center of care in Mexico city.

DETAILED DESCRIPTION:
This is an open label, randomized, prospective clinical trial, with a 1:1:1 aleatorization of a single third level specialized neurological center.

Primary objective: To evaluate the clinical impact of the use of buccal midazolam as a treatment of seizure clusters in comparison with orodispersable clonazepam vs usual care.

Secondary objective: To identify patients that present seizure clusters and risk factors associated with the diagnosis. To evaluate the quality of life after drug administration, to evaluate the adverse events associated with the medications. To establish seizure recurrence and mortality in 6 months' follow up.

ELIGIBILITY:
Inclusion Criteria:

* At least age of 18
* Patient available for follow-up
* Previous diagnosis of epilepsy
* Patient meets criteria for seizure clusters (3 or more seizures in a period of 24 hours)

Exclusion Criteria:

* Risk factors for epilepsy have been identified and uncontrolled.
* Younger than 18 years olf
* Follow- up in another healthcare unit
* No previous epilepsy diagnosis
* Adequate control of epilepsy
* Patient meets criteria for clinical or electrographic status epilepticus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline seizure frequency comparison using buccal midazolam, orodispersable clonazepam versus usual care efficacy for seizure clusters | 1,3 and 6 months
  Seizure frequency description, using the Engel Score of Seizure Outcomes

SECONDARY OUTCOMES:
Change from baseline seizure recurrence in 6 months | 6 months
  Seizure frequency description, using the Engel Score of Seizure outcomes.
Change from baseline quality of life assessed by the QOLIE-31 from baseline | 6 months
  Quality of life questionnaire: QOLIE-31 (Quality Of Life in Epilepsy version 31) is a standarized epilepsy quality of life measuring tool compared to initial score at recruitment. QOLIE-31 consists of 31 items distributed in 7 areas: preoccupation for seizures, general quality of life, emotional well-being, energy/fatigue, cognitive alterations, medication effects, and social functioning. Final evaluation of the points is ranging from 10 points (worse quality of life) and 50 points (best quality of life).

CONTACTS AND LOCATIONS:
Overall Officials: Elma M Paredes-Aragón, MD, Principal Investigator — National Institute of Neurology and Neurosurgery
Locations (1):
- Instituto Nacional de Neurología y Neurocirugía "Dr. Manuel Velasco Suárez", Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No